CLINICAL TRIAL: NCT06727461
Title: Effects of a Home-based Feeding EnhancEment in Dementia (FEED@Home) Intervention on Hospital Readmissions: A Multicenter Randomized Controlled Trial
Brief Title: Effects of FEED@Home Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUEN Jacqueline Kwan Yuk, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21223191
Record Dates: First submitted 2024-06-03; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dementia; Dementia Severe
Keywords: Advanced dementia; Careful hand feeding; Feeding difficulties
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a single-blinded multicenter randomized controlled trial to evaluate the effects of the FEED@home intervention.
  Each patient-family dyad will be randomized in a 1:1 ratio to FEED@home program vs. usual care after completing the baseline interview. Allocation sequence will be generated by a computer program using random block sizes of 4, 8 and 12. The sequence will be put in sequentially numbered opaque sealed envelopes to ensure concealment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Feeding EnhancEment in Dementia (Feed@home) (Experimental): 1. Within 3 days after discharge, a nurse will conduct a teleconsultation (30-45 minutes) with the caregiver to assess feeding issues, and offer recommendations and caregiver education materials on feeding strategies.
  2. In Weeks 1-3 after discharge, there will be 2 home visits by speech therapists (each time 45 - 60 minutes) to assess feeding issues at home and provide instructions on feeding techniques and training.
  3. In week 4, there will be a teleconsultation with the nurse (30 - 45 minutes) to discuss any problems arising.
  4. In Weeks 5-8 after discharge, there will be a home visit by nurse (45 - 60 minutes), followed by a teleconsultation with the nurse in the final week (30 - 45 minutes). An additional visit by the speech therapist may be arranged if needed.
  5. The intervention will be resumed after any pauses resulting from patient readmissions to the hospital.
  Interventions: Other: Home-based Feeding EnhancEment in Dementia (Feed@home)
- Control (No Intervention): The patient will receive usual care from the hospital and follow-up care as instructed by the hospital.

INTERVENTIONS:
Other: Home-based Feeding EnhancEment in Dementia (Feed@home) — The FEED@home program is an 8-week initiative led by a speech therapist (ST) and nurse team through teleconsultations and home visits:
  * Within 3 days after discharge, a nurse teleconsultation with the family caregiver to assess the patient's mealtime behaviors and provide feeding strategy recommendations and educational materials.
  * Two to three home visits by STs during mealtime (depending on the mastery of feeding techniques) to assess swallowing and cognitive feeding issues, providing tailored interventions and proper training of feeding techniques.
  * Two teleconsultations by nurses to assess the caregiver's techniques and provide additional training.
  * One additional home visit during mealtime by a nurse to assess the caregiver's mastery of the feeding techniques through observation.
  * The program lasts 8 weeks, regardless of readmissions, unless the patient converts to tube feeding, moves to a care home, passes away, or withdraws from study.
  Other Names: Feed@home program
  Arms: Home-based Feeding EnhancEment in Dementia (Feed@home)

SUMMARY:
The main goal of this single-blinded multicenter randomized trial is to learn if the 8-week home-based Feeding EnhancEment in Dementia program (FEED@home) works to improve unplanned hospital utilization of advanced dementia patients with feeding problems who reside at home after discharge from hospital. It will also investigate the effect of Feed@home program on outcomes including feeding problem-related readmissions, sustainability on oral feeding, feeding difficulty, malnutrition risk, quality of life of patients with dementia, caregiver satisfaction with care, and caregiver burden.

The questions it aims to answer are:

* Does Feed@home intervention reduce unplanned all-cause hospital readmissions of advanced dementia patients with feeding problems at 1, 2, 3, and 6 months after discharge from the hospital?
* Does Feed@home intervention improve the outcomes including feeding problem-related readmissions, sustainability on oral feeding, feeding difficulty, malnutrition risk, quality of life of patients with dementia, caregiver satisfaction, and burden with care?

Investigators will compare Feed@home intervention to usual care after discharge to see if the Feed@home program improves the outcomes of patients and caregivers. The Feed@home program includes an 8-week follow-up care by speech therapists and nurses via home visits and teleconsultations.

Participants will be dyads of patients and their caregivers, and they will:

* Receive Feed@home intervention or usual care after discharge
* Give consent for access to patients' information and hospital records
* Caregivers to complete questionnaire at recruitment and 2 and 6 months after discharge

DETAILED DESCRIPTION:
To improve in-home post-discharge management of feeding difficulties in advanced dementia patients, our research team members developed the FEED@home intervention with the goals of reducing potentially avoidable hospital readmissions and improving quality of life of advanced dementia patients with feeding difficulties.

This Feed@home intervention was based on existing experience in leading hospital careful hand feeding programs in Hong Kong and a pilot study on the Feeding EnhancEment in Dementia (FEED) program which consists of a hospital-based multidisciplinary intervention and two post-discharge outpatient visits with a speech therapist.

Informed by those experiences, post-discharge follow-up can be enhanced as a hybrid in-home and teleconsultation support service delivered by a speech therapist and nurse team to enable timely support to dementia patients and family caregivers in the home environment post discharge.

We hypothesize that FEED@home can significantly reduce unplanned all-cause and feeding problem-related hospital readmissions, prolong sustainability on oral feeding, reduce feeding difficulty, lessen malnutrition risk, improve quality of life of patients, improve family caregiver satisfaction, and alleviate their care burden.

ELIGIBILITY:
Subjects are dyads of dementia patients and family caregivers.

Inclusion Criteria (For patients):

* Age ≥ 60 years old
* Diagnosis of dementia based on DSM-5 Criteria for Major Neurocognitive Disorder
* Moderately severe to severe dementia as defined by Stage 6 or above on the Functional Assessment Staging Test
* Has indication for tube feeding due to severe feeding difficulties identified by the medical team (cognitive feeding issues and/or oropharyngeal dysphagia) and family surrogate opted for oral feeding
* Maintained on oral feeding at the time of discharge
* Reside at home after discharge
* Has available legally authorized representative (e.g. next of kin) who can provide informed consent for patient

Exclusion Criteria(For patients):

* Any type of feeding tube at time of discharge
* Discharged to residential care homes, respite care or hospice facilities
* No available family caregiver at home

Inclusion Criteria (For family caregivers ):

* Age ≥ 18 years old or above
* Main caregiver who provides or supervises feeding assistance to the patient for ≥70% of meals
* Able to provide informed consent

Exclusion Criteria (For family caregivers ): No specific exclusion criteria

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of unplanned all-cause hospital readmissions | 6-month
  The total number of unplanned all-cause hospital readmissions within the specified time frame will be obtained from electronical medical system. Family caregivers will report any unplanned admissions to private hospitals during the study period.

SECONDARY OUTCOMES:
Number of unplanned all-cause hospital readmissions | 1-month, 2-month, and 3-month
  The total number of unplanned all-cause hospital readmissions within the specified time frame will be obtained from electronical medical system. Family caregivers will report any unplanned admissions to private hospitals during the study period.
Time to first unplanned all-cause hospital readmission | 1-month, 2-month, 3-month and 6-month
  The date of first hospital readmission will be obtained based on a review of medical records. The time from discharge date to the date of first all-cause hospital readmission will be calculated.
Number of unplanned feeding-mode related hospital readmissions | 1-month, 2-month, 3-month and 6-month
  The total number of unplanned feeding mode related hospital readmissions within the specified time frame will be obtained from electronic medical system. Family caregivers will report any unplanned admissions to private hospitals related to feeding mode during the study period.
Time to first unplanned feeding mode related hospital readmission | 1-month, 2-month, 3-month and 6-month
  The time from discharge to the first hospital readmission related to feeding mode will be documented, including the specific date of readmission.
Time to conversion to tube feeding | 6-month
  The time to conversion to tube feeding will be counted from the discharge date to the date of feeding tube insertion within 6 months, which reflects the sustainability of oral feeding. The timing of feeding tube insertion will be recorded based on a review of medical records.
Edinburgh Feeding Evaluation in Dementia Questionnaire-Chinese version (C-EdFED-Q) | Baseline, 2-month, and 6-month
  C-EdFED-Q will assess the patient's feeding difficulty by caregiver's rating of observable feeding behaviors at mealtimes (11 items rated on a 3-point scale from 1 'never' to 2 'often,' score range 0-20; 20=highest difficulty). The C-EdFED-Q has been shown to have good interrater reliability, internal consistency, and construct validity.
Mini Nutritional Assessment-Short Form (MNA-SF) | Baseline, 2-month, 6-month
  MNA-SF assess the malnutrition risk of patients by interviewing the family caregiver. The MNA-SF is a validated 6-item tool for assessing malnutrition in older adults including Chinese patients.24-25 The items assess food intake, unintended weight loss, mobility, acute disease, neuropsychological problems, and BMI or calf circumstance if BMI is unavailable (range 0-14 points, <7 points indicates a state of malnutrition, 7 to 11 at risk of malnutrition, > 11 normal nutritional status)
Quality of Life in Late-Stage Dementia Scale-Chinese version (QUALID-C) | Baseline, 2-month, and 6-month
  QUALID-C will assess the quality of life of patients with advanced dementia. The QUALID-C is a validated 11-item scale rated on a 5-point Likert scale based on caregivers report of observable behaviors of people with severe dementia (range 11-55; lower score indicates higher QoL). The QUALID-C has demonstrated excellent reliability, internal consistency, and validity.
Satisfaction with Care Questionnaire | Baseline, 2-month, and 6-month
  Satisfaction with Care Questionnaire is modified from the questionnaire developed by the Hospital Authority Quality and Safety Subcommittee to assess family caregivers' satisfaction with care services provided to support careful hand feeding (Reference Manual). The 7-item questionnaire is rated on a 5-point Likert scale (1=strongly disagree; 5=strongly agree.
Zarit Burden Interview Scale-Cantonese version (CZBI) | Baseline, 2-month, and 6-month
  This scale will assess caregiver burden by interviewing the family caregiver. The 12-item CZBI-Short is rated on a 5-point Likert scale and has been demonstrated to be a reliable and valid instrument to assess burden in Chinese dementia caregivers

OTHER OUTCOMES:
Qualitative interview | 6-month
  Approximately 15 to 20 family caregivers who have completed the FEED@home intervention, and the speech therapists and nurses involved in the consultation and home visits will be interviewed to understand their perceptions related to the acceptability, feasibility and experience of the FEED@home intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Yuen, M.D., Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be collected and stored confidentially. Electronic data files will be password-protected in encrypted storage devices. Paper data files will be kept in secure file cabinets in a locked office at the study sites. Access to files will be restricted to key study personnel and supervised by the principal investigator of the study.
  There is no plan for IPD sharing.

REFERENCES:
- [Background] Mitchell SL, Teno JM, Kiely DK, Shaffer ML, Jones RN, Prigerson HG, Volicer L, Givens JL, Hamel MB. The clinical course of advanced dementia. N Engl J Med. 2009 Oct 15;361(16):1529-38. doi: 10.1056/NEJMoa0902234. PMID 19828530
- [Background] Cintra MT, de Rezende NA, de Moraes EN, Cunha LC, da Gama Torres HO. A comparison of survival, pneumonia, and hospitalization in patients with advanced dementia and dysphagia receiving either oral or enteral nutrition. J Nutr Health Aging. 2014 Dec;18(10):894-9. doi: 10.1007/s12603-014-0487-3. PMID 25470805
- [Background] Chou HH, Tsou MT, Hwang LC. Nasogastric tube feeding versus assisted hand feeding in-home healthcare older adults with severe dementia in Taiwan: a prognosis comparison. BMC Geriatr. 2020 Feb 14;20(1):60. doi: 10.1186/s12877-020-1464-9. PMID 32059646
- [Background] Kelly S, Lafortune L, Hart N, Cowan K, Fenton M, Brayne C; Dementia Priority Setting Partnership. Dementia priority setting partnership with the James Lind Alliance: using patient and public involvement and the evidence base to inform the research agenda. Age Ageing. 2015 Nov;44(6):985-93. doi: 10.1093/ageing/afv143. PMID 26504119
- [Background] Finucane TE, Christmas C, Travis K. Tube feeding in patients with advanced dementia: a review of the evidence. JAMA. 1999 Oct 13;282(14):1365-70. doi: 10.1001/jama.282.14.1365. PMID 10527184
- [Background] Davies N, Barrado-Martin Y, Vickerstaff V, Rait G, Fukui A, Candy B, Smith CH, Manthorpe J, Moore KJ, Sampson EL. Enteral tube feeding for people with severe dementia. Cochrane Database Syst Rev. 2021 Aug 13;8(8):CD013503. doi: 10.1002/14651858.CD013503.pub2. PMID 34387363
- [Background] Lee YF, Hsu TW, Liang CS, Yeh TC, Chen TY, Chen NC, Chu CS. The Efficacy and Safety of Tube Feeding in Advanced Dementia Patients: A Systemic Review and Meta-Analysis Study. J Am Med Dir Assoc. 2021 Feb;22(2):357-363. doi: 10.1016/j.jamda.2020.06.035. Epub 2020 Jul 29. PMID 32736992
- [Background] DiBartolo MC. Careful hand feeding: a reasonable alternative to PEG tube placement in individuals with dementia. J Gerontol Nurs. 2006 May;32(5):25-33; quiz 34-5. doi: 10.3928/00989134-20060501-06. PMID 16708981
- [Background] Luk JKH, Chan TC, Chan FHW. Letter to the Editor: Careful hand feeding program in a geriatric step-down hospital in Hong Kong - is this feasible? J Frailty Aging. 2021;10(3):303-304. doi: 10.14283/jfa.2020.50. No abstract available. PMID 34105718
- [Background] Yuen JK, Chan FHW, Chan TC, Chow DTY, Chu ST, Shea YF, Luk JKH. Hospital Careful Hand Feeding Program Reduced Feeding Tube Use in Patients with Advanced Dementia. J Nutr Health Aging. 2023;27(6):432-437. doi: 10.1007/s12603-023-1926-9. PMID 37357327
- [Background] Yuen JK, Luk JKH, Chan TC, Shea YF, Chu ST, Bernacki R, Chow DTY, Chan FHW. Reduced Pneumonia Risk in Advanced Dementia Patients on Careful Hand Feeding Compared With Nasogastric Tube Feeding. J Am Med Dir Assoc. 2022 Sep;23(9):1541-1547.e2. doi: 10.1016/j.jamda.2022.03.011. Epub 2022 Apr 27. PMID 35489380